CLINICAL TRIAL: NCT00145717
Title: China Plant Sterol Trial - A Randomised Trial to Determine the Effects on Blood Cholesterol Levels of a Milk Tea Product Enriched With Plant Sterol Among 300 Chinese Living in Beijing
Brief Title: China Plant Sterol Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: Peking University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CPST
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2005-09-05 (Estimated); Status verified 2005-09

CONDITIONS: Hypercholesterolemia; Cardiovascular Diseases
Keywords: Phytosterols; Cholesterol; China; Randomized controlled trial
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases

INTERVENTIONS:
Drug: Plant sterol enriched milk tea

SUMMARY:
The aim of this study is to see if plant sterols are effective at lowering blood cholesterol levels in Chinese people. The study will be done with Chinese colleagues based at Peking University in Beijing with whom our Institute has a well-established collaboration. The study will be randomised, placebo-controlled and double-blind. The total study period for participants will be an average of seven weeks comprised of a two-week placebo run-in period and a five-week follow-up on randomised treatment. Randomised treatment will comprise either placebo, low- or standard-dose plant sterol. The primary outcome for the study will be blood cholesterol levels.

DETAILED DESCRIPTION:
RESEARCH PLAN The study is a randomised, double-blind, placebo-controlled trial with three parallel groups, two assigned different doses of active treatment and one assigned placebo. The total study period for participants will be an average of seven weeks comprised of a two-week placebo treatment run-in period prior to randomisation and a five-week follow-up on randomised treatment. An estimated 400 participants will be commenced on run-in with the expectation that 300 (100 in each group) will go on to randomisation.

STUDY TREATMENTS Pre-randomisation open run-in phase: All potentially eligible participants will commence a 10-20 days run-in period with the placebo milk tea administered twice daily. This run-in period will help to identify before randomisation, those individuals who are unlikely to tolerate the milk tea product or comply with the study follow up procedures.

Post randomisation double-blind treatment phase: Participants that successfully complete the run-in phase will be assigned at random to receive either:

* Milk tea containing a total of 2.3g of plant sterol each day administered in two divided doses of 1.15g; or
* Milk tea containing a total of 1.5g of plant sterol each day administered in two divided doses of 0.75g; or
* Placebo milk tea containing no plant sterol. Blinding of participants and investigators will be assured by providing all groups with their allocated treatment in packaging that is identical except for a unique identifying number corresponding to the randomisation code.

Comparisions:

* 2.3g/d treatment group compared to placebo group
* 1.5g/d treatment group compared to placebo group
* active treatment group (2.3g/d and 1.5g/d combined) compared to placebo group
* 2.3g/d treatment group compared to 1.5g/d treatment group
* Secondary: To establish the effects of the same intervention on total cholesterol levels.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria will be:

* Age between 18 and 65 years old (inclusive) at baseline
* Able to provide informed consent
* Usual diet that includes significant fat consumption at the main meals eaten each week and/or a history of hypercholesterolemia
* Participant is likely to comply with the study treatment during the study period

Exclusion Criteria:

Participants will be excluded on the basis of:

* Known serious gastrointestinal disease or other serious illness. Individuals with stable cardiovascular disease will, however, be eligible
* Known lactose intolerance or diet that excludes dairy products
* Known Sitosterolaemia (a very rare genetic condition causing very high blood sitosterol levels)
* Current hospitalisation
* Current use of drug with likely significant impact on gastro-intestinal absorption of cholesterol or plant sterol (e.g. ezetimibe, bile acid-binding resins, or orlistat)
* Participant is currently using or is planning to use non-trial plant sterol/stanol-containing products for the seven week study period
* Participation in another study within last 3 months
* Pregnant or planning to become pregnant in next three months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-04; Study Completion 2005-07

PRIMARY OUTCOMES:
Low density lipoprotein cholesterol levels

SECONDARY OUTCOMES:
Total cholesterol levels;
High density lipoprotein cholesterol levels;
Triglycerides levels;
Liking and adherence

CONTACTS AND LOCATIONS:
Overall Officials: Bruce C Neal, MRCP, PhD, Principal Investigator — The George Institute
Locations (1):
- Peking University Health Science Centre, Beijing, China

REFERENCES:
- [Derived] Li NY, Li K, Qi Z, Demonty I, Gordon M, Francis L, Molhuizen HO, Neal BC. Plant sterol-enriched milk tea decreases blood cholesterol concentrations in Chinese adults: a randomised controlled trial. Br J Nutr. 2007 Nov;98(5):978-83. doi: 10.1017/S0007114507754302. Epub 2007 Jul 9. PMID 17617940